CLINICAL TRIAL: NCT02690883
Title: Effect of Exenatide on 24h-UAER in Patients With Diabetic Nephropathy: a 24- Week Study
Brief Title: Effect of Exenatide on 24h-UAER in Patients With Diabetic Nephropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Yaoming Xue, Department of Endocrinology and Metabolism, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ESR-14-10425
Record Dates: First submitted 2016-02-20; First posted 2016-02-24 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Diabetic Nephropathies
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Exenatide; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lispro (Active Comparator): Patients are treated with Glargine (Lantus, Sanofi-Aventis), the dosage is initiated according to the previous treatment plan and weight of the patients, injection before bed time, titration following FPG <7.2mmol/L and >4.4mmol/L.
  Interventions: Drug: Lispro
- Exenatide (Experimental): Patients are treated with Glargine (Lantus, Sanofi-Aventis), the dosage is initiated according to the previous treatment plan and weight of the patients, injection before bed time, titration following FPG <7.2mmol/L and >4.4mmol/L.
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Exenatide — Exenatide (Astrazeneca ) 5 μg(initial dose)/10ug(maintenance dose) Subcutaneous injection Bid
  Other Names: Byetta
  Arms: Exenatide
Drug: Lispro — Lispro (Eli Lilly), the dosage is initiated according to the previous treatment plan and weight of the patients, distribute the dosage to 1:1:1 before 3 meals, titration following PPG <10.0mmol/L.
  Other Names: Humalog
  Arms: Lispro

SUMMARY:
This is a multi-center, randomized, parallel study to evaluate effect of exenatide on 24h-UAER in patients with diabetic nephropathy.

Screening will be made to select eligible participants before intervention. The trial will include 2-week run-in period of stable doses of glargine plus lispro insulin and 24-week treatment period. After the run-in period, patients were randomly assigned to one of two groups for antihyperglycaemic therapies for a total of 24-weeks: glargine plus exenatide and continued glargine plus lispro insulin. The treatment of exenatide will be initiated by 5ug bid, and uptitrated to 10 ug bid after 4 weeks and then maintained at 10ug bid until the completion of the study. Lispro insulin will be initially treated according to the insulin dosage of previous antihyperglycaemic therapies, and further titrated up at 4-week intervals until to reach the target fasting blood glucose (FPG).

DETAILED DESCRIPTION:
Objective:

To evaluate effect of exenatide on 24-UAER in patients with diabetic nephropathy

Hypothesis:

Compared with glargine plus lispro group, at 24 weeks, glargine plus exenatide group can: 1) take more significant reduction of 24h-UAER; 2) take more reduction of ACR; 3) take more weight loss, blood pressure reduction; 4) take lower hypoglycemia incidence and less insulin dosage.

Primary endpoint： The proportion of reduction of 24h-UAER(urinary albumin excretion rates)

Secondary endpoints： 24h-UAER at 24 weeks; the rate of urinary albumin to creatinine ratio(ACR) change at 24 weeks; HbA1c, FPG,PPG, weight , BP

Treatment duration： 24weeks

Patient/Sites： 90 patients / 3 sites

Timeline (best case)： Planed duration of recruitment period: 6 month Planed date for first screening: 1 October 2015 Planed completion of the last subject: 1 March 2017 Planned completion of clinical trial report: 30 October 2017

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures.
2. Diagnosed with type 2 diabetes with HbA1c ≥ 7.0% and ≤ 11.0% at screening (the result is valid for seven days).
3. Men and women (non-pregnant and using a medically approved birth-control method) aged from 18 to 80 at screening.
4. Body mass index (BMI) ≥18 and ≤35 kg/m2.
5. Blood Pressure (BP) ≥ 90/60mmHg and ≤160/100mmHg.

6.24h urinary albumin excretion rate (UAE) >0.3g/24h after 3 months treatment with several hypoglycemic agents (sulphonylureas, metformin, AG-inhibitor, meglitinides or insulin), ACEI/ARB and salt restriction(the result is valid for seven days).

7.eGFR >30ml/min(the result is valid for seven days).

Exclusion Criteria:

1．Women who are pregnant, intending to become pregnant during the study period, currently lactating females, or women of child-bearing potential not using highly effective, medically approved birth control methods.

2. Diagnosis or history of:

1. Type 1 diabetes mellitus, diabetes resulting from pancreatic injury or secondary forms of diabetes, eg, acromegaly or Cushing's syndrome.
2. Acute metabolic diabetic complications such as ketoacidosis or hyperosmolar coma within the past 6 months.

   3. Previous treatment with any Thiazolidinediones (TZDs), dipeptidyl peptidase-4 (DPP4) inhibitor or GLP-1 receptor agonists within the past 3 months.

   4. History of hypersensitivity reaction (e.g., anaphylaxis, angioedema, exfoliative skin conditions) to exenatide.

   5. Blood amylase and/or lipase > 2 times the upper limit of the normal (ULN) laboratory range.

   6. Hyperkalemia (K+>5.5mmol/L).

   7. eGFR <30ml/min/1.73m2.

   8. Patients without diabetic retinopathy.

   9. Triglycerides (fasting) > 4.5 mmol/L (400 mg/dL) at screening or within 4 weeks prior to screening (by local laboratory).

   10. Patients with clinically apparent liver disease characterized by ALT or AST > 3ULN confirmed on two consecutive measurements (by local laboratory) within 4 weeks prior to screening period.

   11. Significant cardiovascular history within the past 3 months prior to screening defined as: myocardial infarction, coronary angioplasty or bypass graft(s), valvular disease or repair, unstable angina pectoris, transient ischemic attack, or cerebrovascular accident.

   12. Congestive heart failure defined as New York Heart Association (NYHA) class III or IV.

   13. History of chronic pancreatitis or idiopathic acute pancreatitis.

   14. History of medullary thyroid carcinoma.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2016-04-08 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
the percentage change of 24h-UAER(urinary albumin excretion rates) from baseline at Week 24 | from baseline at Week 24
  the percentage change of 24h-UAER=(24h-UAERweek24 - 24h-UAERbaseline)/ 24h-UAERbaseline

SECONDARY OUTCOMES:
the percentage change of ACR | from baseline at Week 24
  the percentage change of ACR=(ACRweek24 - ACRbaseline)/ ACRbaseline
Change in 24h-UAER | from baseline at Week 24
  Change in 24h-UAER =24h-UAERweek24 - 24h-UAERbaseline
Change in HbA1c | from baseline at Week 24
  Change in HbA1c=HbA1cweek24-HbA1cbaseline
Change in FPG | from baseline at Week 24
  Change in FPG=FPGweek24-FPGbaseline
Change in Weight | from baseline at Week 24
  Change in weight=Weightweek24-Weightbaseline
Change in Blood pressure | from baseline at Week 24
  Change in blood pressure=SBPweek24-SBPbaseline

CONTACTS AND LOCATIONS:
Overall Officials: Xue, PhD, Principal Investigator — Department of Endocrinology & Metabolism, Nanfang Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] KDOQI. KDOQI Clinical Practice Guidelines and Clinical Practice Recommendations for Diabetes and Chronic Kidney Disease. Am J Kidney Dis. 2007 Feb;49(2 Suppl 2):S12-154. doi: 10.1053/j.ajkd.2006.12.005. No abstract available. PMID 17276798
- [Background] Lim AKh. Diabetic nephropathy - complications and treatment. Int J Nephrol Renovasc Dis. 2014 Oct 15;7:361-81. doi: 10.2147/IJNRD.S40172. eCollection 2014. PMID 25342915
- [Background] de Zeeuw D, Parving HH, Henning RH. Microalbuminuria as an early marker for cardiovascular disease. J Am Soc Nephrol. 2006 Aug;17(8):2100-5. doi: 10.1681/ASN.2006050517. Epub 2006 Jul 6. PMID 16825327
- [Background] Filippatos TD, Elisaf MS. Effects of glucagon-like peptide-1 receptor agonists on renal function. World J Diabetes. 2013 Oct 15;4(5):190-201. doi: 10.4239/wjd.v4.i5.190. PMID 24147203
- [Background] Lu B, Song X, Dong X, Yang Y, Zhang Z, Wen J, Li Y, Zhou L, Zhao N, Zhu X, Hu R. High prevalence of chronic kidney disease in population-based patients diagnosed with type 2 diabetes in downtown Shanghai. J Diabetes Complications. 2008 Mar-Apr;22(2):96-103. doi: 10.1016/j.jdiacomp.2007.08.001. PMID 18280439
- [Background] Lai X, Zhang AH, Chen SY, He L, Su CY, Fan MH, Wang T. Outcomes of stage 1-5 chronic kidney disease in Mainland China. Ren Fail. 2014 May;36(4):520-5. doi: 10.3109/0886022X.2013.875859. Epub 2014 Jan 23. PMID 24456114
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Tomino Y. Pathogenesis and treatment of chronic kidney disease: a review of our recent basic and clinical data. Kidney Blood Press Res. 2014;39(5):450-89. doi: 10.1159/000368458. Epub 2014 Nov 30. PMID 25501571
- [Background] Kobori H, Mori H, Masaki T, Nishiyama A. Angiotensin II blockade and renal protection. Curr Pharm Des. 2013;19(17):3033-42. doi: 10.2174/1381612811319170009. PMID 23176216
- [Background] Park CW, Kim HW, Ko SH, Lim JH, Ryu GR, Chung HW, Han SW, Shin SJ, Bang BK, Breyer MD, Chang YS. Long-term treatment of glucagon-like peptide-1 analog exendin-4 ameliorates diabetic nephropathy through improving metabolic anomalies in db/db mice. J Am Soc Nephrol. 2007 Apr;18(4):1227-38. doi: 10.1681/ASN.2006070778. Epub 2007 Mar 14. PMID 17360951
- [Background] Xu WW, Guan MP, Zheng ZJ, Gao F, Zeng YM, Qin Y, Xue YM. Exendin-4 alleviates high glucose-induced rat mesangial cell dysfunction through the AMPK pathway. Cell Physiol Biochem. 2014;33(2):423-32. doi: 10.1159/000358623. Epub 2014 Feb 11. PMID 24556697
- [Background] Zhang H, Zhang X, Hu C, Lu W. Exenatide reduces urinary transforming growth factor-beta1 and type IV collagen excretion in patients with type 2 diabetes and microalbuminuria. Kidney Blood Press Res. 2012;35(6):483-8. doi: 10.1159/000337929. Epub 2012 Jun 8. PMID 22687869
- [Background] Imamura S, Hirai K, Hirai A. The glucagon-like peptide-1 receptor agonist, liraglutide, attenuates the progression of overt diabetic nephropathy in type 2 diabetic patients. Tohoku J Exp Med. 2013 Sep;231(1):57-61. doi: 10.1620/tjem.231.57. PMID 24064677
- [Background] Ahmad SR, Swann J. Exenatide and rare adverse events. N Engl J Med. 2008 May 1;358(18):1970-1; discussion 1971-2. No abstract available. PMID 18456920
- [Background] Bloomgren G, Braum D, Kolterman O. Exenatide and rare adverse events. N Engl J med 2008; 358: 1971-2.
- [Background] Yanagisawa K, Ashihara J, Obara S, Wada N, Takeuchi M, Nishino Y, Maeda S, Ishibashi Y, Yamagishi S. Switching to multiple daily injection therapy with glulisine improves glycaemic control, vascular damage and treatment satisfaction in basal insulin glargine-injected diabetic patients. Diabetes Metab Res Rev. 2014 Nov;30(8):693-700. doi: 10.1002/dmrr.2537. PMID 24639403
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952